CLINICAL TRIAL: NCT05274841
Title: Implementation of Systematic Support of Relatives of Palliative Care Patients : a Cohort Study
Brief Title: Systematic Support for Relatives of Palliative Care Patients
Acronym: BALANCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Julie Høgh Rasmussen, Psychologist, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P-2020-429
Record Dates: First submitted 2022-01-28; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Prolonged Grief Disorder
Keywords: Palliative Care; Screening tool; Assessment tool; Relatives; Support needs; Anticipatory Grief; Palliative patients; Caregivers
MeSH Terms: conditions — Prolonged Grief Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Identified support needs (Other): Identified need of either support from a psychologist, nurse, doctor, socialworker or a combination of theese.
  Interventions: Other: Support of relatives

INTERVENTIONS:
Other: Support of relatives — Screening of the support needs of relatives

SUMMARY:
The primary purpose of this study is to validate the prognostic screening tool from The Aarhus Bereavement Study (TABS) and to implement a systematic support for relatives of palliative care patients in order to prevent the development of prolonged grief disorder. Depending on their identified support needs, the relatives are offered different interventions. It is evaluated whether this procedure of screening and intervening are able to reduce the risk of developing prolonged grief disorder.

DETAILED DESCRIPTION:
PRIMARY OUTCOME: identification of the support needs of relatives of palliative care patients

SECONDARY OUTCOME: evaluation of the initiated interventions and whether these are able to reduce the risk of developing prolonged grief disorder

PARTICIPANTS: Relatives (age 18-90) of patients affiliated with specialized palliative care in The Capital Region of Denmark.

The relatives will complete a survey and prognostic screening tool at respectively 2 weeks (T1) and every 6 months (T2) from the time that the patients is affiliated to the specialized palliative care and until the death of the patient. This will happen regardless the status of the patient - that is, whether or not the patient continues being affiliated with specialized palliative care, or the patient is being referred to another palliative care units or doesn't need palliative care anymore.

Furthermore the relatives will complete a follow-up survey and the diagnostic questionnaire PGD-13 at respectively 6 months (T3) and 18 months (T4) after the death of the patient (post loss). It will be evaluated whether there are any diffences in the grief symptoms of relatives of patients with a malign versus non-malign disease. It will also be evaluated whether there is an association between the intervention the relatives received from the palliative care unit at Rigshospital and their grief symptoms post loss.

ELIGIBILITY:
Inclusion Criteria:

* relatives of palliative care patients with relation to Department of Palliative Care, (Rigshospitalet)
* relatives identified by the patient

Exclusion Criteria:

* relatives who do not read or understand danish
* relatives who are cognitive disabled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Support needs of relatives of palliative patients (baseline) | 1 month from the time that the patient is referred to the palliative care team.
  Identification of support needs of relatives assessed by the prognostic screening tool from The Aarhus Bereavement Study (TABS).
Change in Support needs of relatives of palliative patients from baseline | 6 months
  Identification of support needs of relatives assessed by the prognostic screening tool from
Change in Support needs of relatives of palliative patients from baseline | 12 months
  Identification of support needs of relatives assessed by the prognostic screening tool from
Change in Support needs of relatives of palliative patients from baseline | 18 months
  Identification of support needs of relatives assessed by the prognostic screening tool from

SECONDARY OUTCOMES:
Prolonged grief | 6 months post-loss.
  Symptoms of prolonged grief measured using the Prolonged Grief Disorder - 13 (PG-13, Prigerson et al, 2009). Scores ranging from 11 to 55 are used in the current study, and a higher score indicates a worse outcome. However, there are no officially recommended cut-off scores (Pohlkamp et al, 2018).
Prolonged grief | 18 months post-loss.
  Symptoms of prolonged grief measured using the Prolonged Grief Disorder - 13 (PG-13, Prigerson et al, 2009). Scores ranging from 11 to 55 are used in the current study, and a higher score indicates a worse outcome. However, there are no officially recommended cut-off scores (Pohlkamp et al, 2018).

CONTACTS AND LOCATIONS:
Locations (1):
- Julie Høgh Rasmussen, Copenhagen, Vesterbro, Denmark

IPD SHARING:
Plan to Share IPD: No